CLINICAL TRIAL: NCT06328738
Title: A Phase 1a/1b Study of ELVN-002 Combined With Trastuzumab in Advanced Stage HER2+ Solid Tumors, and ELVN-002 Combined With Trastuzumab and Chemotherapy in Advanced Stage HER2+ Colorectal Cancer and Breast Cancer
Brief Title: ELVN-002 With Trastuzumab +/- Chemotherapy in HER2+ Solid Tumors, Colorectal and Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Enliven Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ELVN-002-003
Record Dates: First submitted 2024-03-10; First posted 2024-03-25 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-07

CONDITIONS: HER2-positive Breast Cancer; HER2-positive Gastric Cancer; HER2 Positive Solid Tumors; HER2 Amplification; Colorectal Cancer
Keywords: ELVN-002; HER2 positive Colorectal Cancer; HER2 overexpression; HER2
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Trastuzumab; Fluorouracil; Oxaliplatin; Capecitabine; eribulin; Paclitaxel; Leucovorin

STUDY DESIGN:
Intervention Model Description: Phase 1a will be a dose escalation of ELVN-002 in combination with fixed doses of trastuzumab or trastuzumab + chemotherapy according to the Bayesian Optimal Interval Design model. Phase 1b will be a dose expansion at one or more doses of ELVN-002.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Part 1: ELVN-002 + trastuzumab dose escalation (Experimental): ELVN-002 will be administered by mouth (orally) once or twice a day from cycle 1 day 1 onwards. Trastuzumab will be administered IV (intravenously) in 21-day cycles, at 8mg/kg on cycle 1 day 2 followed by a dose of 6mg/kg on day 1 of cycles 2+.
  Interventions: Drug: ELVN-002; Drug: Trastuzumab
- Part 2A: ELVN-002 + trastuzumab + CAPEOX dose escalation in colorectal cancer (Experimental): ELVN-002 will be administered by mouth (orally) once or twice a day from cycle 1 day 1 onwards. Trastuzumab will be administered IV (intravenously) in 21-day cycles, at 8mg/kg on cycle 1 day 2 followed by a dose of 6mg/kg on day 1 of cycles 2+. Capecitabine will be administered orally twice daily at 1000 mg/m2 on days 1 - 14 of a 21-day cycle. Oxaliplatin will be administered intravenously at 130 mg/m2 on day 1 of a 21-day cycle.
  Interventions: Drug: ELVN-002; Drug: Trastuzumab; Drug: Oxaliplatin; Drug: Capecitabine
- Part 2B: ELVN-002 + trastuzumab + mFOLFOX6 dose escalation in colorectal cancer (Experimental): ELVN-002 will be administered by mouth (orally) once or twice a day from cycle 1 day 1 onwards. Trastuzumab will be administered intravenously at 6 mg/kg IV cycle 1, day 2 followed by 4 mg/kg IV cycle 1, day 15, and then one dose at 4mg/kg IV every 14 days. Fluorouracil (5-FU) will be administered intravenously as a 400 mg/m2 IV bolus on days 1 and 15 followed by 2400 mg/m2 over 46-48 hours of continuous infusion on days 1-3 and days 15-17 of a 28-day cycle. Leucovorin will be administered intravenously at 400 mg/m2 concurrently with oxaliplatin on days 1 and 15 of a 28-day cycle. Oxaliplatin will be administered intravenously at 85 mg/m2 IV on day 1 and 15 of a 28-day cycle.
  Interventions: Drug: ELVN-002; Drug: Trastuzumab; Drug: 5-Fluorouracil; Drug: Oxaliplatin; Drug: Leucovorin
- Part 2C: ELVN-002 + trastuzumab + capecitabine dose escalation in breast cancer (Experimental): ELVN-002 will be administered by mouth (orally) once or twice a day from cycle 1 day 1 onwards. Trastuzumab will be administered IV (intravenously) in 21-day cycles, at 8mg/kg on cycle 1 day 2 followed by a dose of 6mg/kg on day 1 of cycles 2+. Capecitabine will be administered orally twice daily at 1000 mg/m2 on days 1 - 14 of a 21-day cycle.
  Interventions: Drug: ELVN-002; Drug: Trastuzumab; Drug: Capecitabine
- Part 2D: ELVN-002 + trastuzumab + paclitaxel dose escalation in solid tumors (Experimental): ELVN-002 will be administered by mouth (orally) once or twice a day from cycle 1 day 1 onwards. Trastuzumab will be administered IV (intravenously) in 21-day cycles, at 8mg/kg on cycle 1 day 2 followed by a dose of 6mg/kg on day 1 of cycles 2+. Paclitaxel will be administered intravenously at 80 mg/m2 on days 1, 8, and 15 of a 21-day cycle.
  Interventions: Drug: ELVN-002; Drug: Trastuzumab; Drug: paclitaxel
- Part 2E: ELVN-002 + trastuzumab + eribulin dose escalation in breast cancer (Experimental): ELVN-002 will be administered by mouth (orally) once or twice a day from cycle 1 day 1 onwards. Trastuzumab will be administered IV (intravenously) in 21-day cycles, at 8mg/kg on cycle 1 day 2 followed by a dose of 6mg/kg on day 1 of cycles 2+. Eribulin will be administered intravenously at 1.4 mg/m2 on days 1 and 8 of a 21-day cycle.
  Interventions: Drug: ELVN-002; Drug: Trastuzumab; Drug: Eribulin
- Part 3A: ELVN-002 + trastuzumab dose expansion in colorectal cancer (Experimental): ELVN-002 will be administered by mouth (orally) once or twice a day from cycle 1 day 1 onwards. Trastuzumab will be administered IV (intravenously) in 21-day cycles, at 8mg/kg on cycle 1 day 2 followed by a dose of 6mg/kg on day 1 of cycles 2+
  Interventions: Drug: ELVN-002; Drug: Trastuzumab
- Part 3B: ELVN-002 + trastuzumab dose expansion in breast cancer (Experimental): ELVN-002 will be administered by mouth (orally) once or twice a day from cycle 1 day 1 onwards. Trastuzumab will be administered IV (intravenously) in 21-day cycles, at 8mg/kg on cycle 1 day 2 followed by a dose of 6mg/kg on day 1 of cycles 2+.
  Interventions: Drug: ELVN-002; Drug: Trastuzumab
- Part 3C: ELVN-002 + trastuzumab dose expansion in other solid tumor type 1 (Experimental): ELVN-002 will be administered by mouth (orally) once or twice a day from cycle 1 day 1 onwards. Trastuzumab will be administered IV (intravenously) in 21-day cycles, at 8mg/kg on cycle 1 day 2 followed by a dose of 6mg/kg on day 1 of cycles 2+.
  Interventions: Drug: ELVN-002; Drug: Trastuzumab
- Part 3D: ELVN-002 + trastuzumab dose expansion in other solid tumor type 2 (Experimental): ELVN-002 will be administered by mouth (orally) once or twice a day from cycle 1 day 1 onwards. Trastuzumab will be administered IV (intravenously) in 21-day cycles, at 8mg/kg on cycle 1 day 2 followed by a dose of 6mg/kg on day 1 of cycles 2+.
  Interventions: Drug: ELVN-002; Drug: Trastuzumab
- Part 3E: ELVN-002 + trastuzumab dose expansion in other solid tumor type 3 (Experimental): ELVN-002 will be administered by mouth (orally) once or twice a day from cycle 1 day 1 onwards. Trastuzumab will be administered IV (intravenously) in 21-day cycles, at 8mg/kg on cycle 1 day 2 followed by a dose of 6mg/kg on day 1 of cycles 2+.
  Interventions: Drug: ELVN-002; Drug: Trastuzumab
- Part 4A: ELVN-002 + trastuzumab + CAPEOX dose expansion in colorectal cancer (Experimental): ELVN-002 will be administered by mouth (orally) once or twice a day from cycle 1 day 1 onwards. Trastuzumab will be administered IV (intravenously) in 21-day cycles, at 8mg/kg on cycle 1 day 2 followed by a dose of 6mg/kg on day 1 of cycles 2+. Capecitabine will be administered orally twice daily at 1000 mg/m2 on Days 1 - 14 of a 21-day cycle. Oxaliplatin: will be administered intravenously at 130 mg/m2 on Day 1 of a 21-day cycle.
  Interventions: Drug: ELVN-002; Drug: Trastuzumab; Drug: Oxaliplatin; Drug: Capecitabine
- Part 4B: ELVN-002 + trastuzumab + mFOLFOX6 dose expansion in colorectal cancer (Experimental): ELVN-002 will be administered by mouth (orally) once or twice a day from cycle 1 day 1 onwards. Trastuzumab will be administered intravenously at 6 mg/kg IV cycle 1, day 2 followed by 4 mg/kg IV cycle 1, day 15, and then one dose at 4mg/kg IV every 14 days. Fluorouracil (5-FU) will be administered intravenously as a 400 mg/m2 IV bolus on days 1 and 15 followed by 2400 mg/m2 over 46-48 hours of continuous infusion on days 1-3 and days 15-17 of a 28-day cycle. Leucovorin will be administered intravenously at 400 mg/m2 concurrently with oxaliplatin on days 1 and 15 of a 28-day cycle. Oxaliplatin will be administered intravenously at 85 mg/m2 IV on days 1 and 15 of a 28-day cycle.
  Interventions: Drug: ELVN-002; Drug: Trastuzumab; Drug: 5-Fluorouracil; Drug: Oxaliplatin; Drug: Leucovorin

INTERVENTIONS:
Drug: ELVN-002 — capsule
Drug: Trastuzumab — intravenous
Drug: 5-Fluorouracil — intravenous
  Arms: Part 2B: ELVN-002 + trastuzumab + mFOLFOX6 dose escalation in colorectal cancer; Part 4B: ELVN-002 + trastuzumab + mFOLFOX6 dose expansion in colorectal cancer
Drug: Oxaliplatin — intravenous
  Arms: Part 2A: ELVN-002 + trastuzumab + CAPEOX dose escalation in colorectal cancer; Part 2B: ELVN-002 + trastuzumab + mFOLFOX6 dose escalation in colorectal cancer; Part 4A: ELVN-002 + trastuzumab + CAPEOX dose expansion in colorectal cancer; Part 4B: ELVN-002 + trastuzumab + mFOLFOX6 dose expansion in colorectal cancer
Drug: Capecitabine — capsule
  Arms: Part 2A: ELVN-002 + trastuzumab + CAPEOX dose escalation in colorectal cancer; Part 2C: ELVN-002 + trastuzumab + capecitabine dose escalation in breast cancer; Part 4A: ELVN-002 + trastuzumab + CAPEOX dose expansion in colorectal cancer
Drug: Eribulin — intravenous
  Arms: Part 2E: ELVN-002 + trastuzumab + eribulin dose escalation in breast cancer
Drug: paclitaxel — intravenous
  Arms: Part 2D: ELVN-002 + trastuzumab + paclitaxel dose escalation in solid tumors
Drug: Leucovorin — intravenous
  Arms: Part 2B: ELVN-002 + trastuzumab + mFOLFOX6 dose escalation in colorectal cancer; Part 4B: ELVN-002 + trastuzumab + mFOLFOX6 dose expansion in colorectal cancer

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and recommended dose of ELVN-002 in combination with trastuzumab in participants with advanced-stage HER2-positive tumors and in combination with trastuzumab, and chemotherapy in participants with advanced-stage HER2-positive colorectal cancer and breast cancer.

DETAILED DESCRIPTION:
Parts 1 and 3 of this study are designed to evaluate preliminary safety, tolerability, and pharmacokinetics (PK) of ELVN-002 in combination with trastuzumab in participants with advanced stage HER2 positive solid tumors. In addition, Part 3 will evaluate the preliminary efficacy of ELVN-002 in combination with trastuzumab in participants with advanced-stage HER2-positive solid tumors.

Part 2 of this study will evaluate the preliminary safety, tolerability, and PK of ELVN-002 in combination with trastuzumab and chemotherapy; capecitabine and oxaliplatin(CAPEOX) or 5-fluorouracil (5-FU), leucovorin (LCV) and oxaliplatin (mFOLFOX6) in participants with advanced stage HER2 positive colorectal cancer, or eribulin or capecitabine in participants with advanced-stage HER2-positive breast cancer, or paclitaxel in participants with advanced stage solid tumors.

In part 4, the preliminary safety, tolerability, PK, and efficacy of ELVN-002 in combination with trastuzumab and CAPEOX or mFOLFOX6 will be evaluated in participants with HER2-positive colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or histologically documented solid tumor.
* Locally advanced or relapsed/refractory disease or unresectable metastatic disease.
* HER2-positive disease based on the following local testing:

  * Colorectal cancer: IHC3+, IHC2+/ISH+, NGS amplification by tissue (no RAS or BRAF mutation allowed)
  * Breast cancer: IHC3+ or IHC2+/ISH+ by tissue
  * Gastric cancer: IHC3+ or IHC2+/ISH+ by tissue
  * Other cancers: IHC3+, IHC2+/ISH+, NGS amplification by tissue or ctDNA
* Prior therapies for Part 1 (Dose Escalation ELVN-002 + trastuzumab):

  * Colorectal cancer: treated with prior fluoropyrimidine, oxaliplatin, irinotecan-based regimens, anti-epidermal growth factor receptor (EGFR) treatment (if clinically indicated), anti-vascular endothelial growth factor (VEGF) treatment (if clinically indicated), and an anti-programmed death ligand 1 (PD-(L)-1) treatment (if the tumor is microsatellite instability (MSI)-high/deficient mismatch repair (dMMR)
  * Breast cancer: treated with prior taxane, pertuzumab, trastuzumab, and fam-trastuzumab deruxtecan (T-DXd) if available and appropriate based on local standard of care and investigator's assessment
  * Gastric cancer: treated with trastuzumab/platinum fluorouracil containing regimen and T-DXd.
  * Other cancers: progressed during or after ≥ 1 prior line of systemic therapy for locally advanced unresectable or metastatic disease
  * Prior HER2 targeted therapy is allowed
* Prior therapies for Part 2 (Phase 1a Dose Escalation ELVN-002 + trastuzumab + chemotherapy):

  * Colorectal cancer: candidate for CAPEOX (capecitabine and oxaliplatin) or mFOLFOX6 (5-FU, LCV and oxaliplatin), and treated, if clinically indicated, with an anti-programmed death ligand 1 (PD-(L)-1) treatment (if the tumor is microsatellite instability (MSI)-high/deficient mismatch repair (dMMR). Prior HER2 targeted therapy is allowed.
  * Breast cancer: candidate for capecitabine, paclitaxel or eribulin, and treated with prior taxane, pertuzumab, trastuzumab, and T-DXd, if available and appropriate, based on local standard of care and investigator's assessment. No prior HER2 targeted tyrosine kinase inhibitor therapy (antibody-drug conjugates and antibodies are allowed), no prior capecitabine (for the capecitabine cohort), no prior eribulin (for the eribulin cohort), and no taxane as immediate prior therapy (paclitaxel cohort).
* Prior therapies for Part 3 (Phase 1b Dose Expansion ELVN-002 + trastuzumab):

  * Colorectal cancer: treated with prior fluoropyrimidine, oxaliplatin, irinotecan-based regimens, anti-epidermal growth factor receptor (EGFR) treatment (if clinically indicated), anti-vascular endothelial growth factor (VEGF) treatment (if clinically indicated), and an anti-programmed death ligand 1 (PD-(L)-1) treatment if the tumor is microsatellite instability (MSI)-high/deficient mismatch repair (dMMR). No prior HER2 targeted therapy.
  * Breast cancer: treated with prior taxane, pertuzumab, trastuzumab, and T-DXd if available and appropriate based on local standard of care and investigator's assessment. No prior HER2 targeted tyrosine kinase inhibitor therapy (antibody-drug conjugates and antibodies are allowed).
  * Gastric cancer: treated with prior trastuzumab/platinum fluorouracil containing regimen and T-DXd. No prior HER2 targeted therapy.
  * Other cancers: Progressed during or after ≥ 1 prior line of systemic therapy for locally advanced unresectable or metastatic disease. No prior HER2 targeted therapy.
* Prior therapies for Part 4 (Phase 1b Dose Expansion ELVN-002 + trastuzumab + chemotherapy):

  * Colorectal cancer: candidate for CAPEOX or mFOLFOX6 and not a candidate for first-line anti-programmed death ligand 1 (PD-(L)-1) treatment (if the tumor is microsatellite instability (MSI)-high/deficient mismatch repair (dMMR). No prior therapy for metastatic disease (1 cycle of mFOLFOX6 or 1 cycle of CAPEOX allowed). No prior HER2 targeted therapy.
* At least 1 measurable lesion based on RECIST v 1.1 within 6 weeks before the first dose of ELVN-002 (Part 3 and Part 4 only; Phase 1b Dose Expansion cohorts)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Adequate hematological, hepatic, renal, and cardiac function

Exclusion Criteria:

* Treatment with anticancer therapy within a specific time before the first dose:

  * Chemotherapy (including ADC) ≤ 3 weeks
  * Immunotherapy ≤ 4 weeks
  * Hormonal therapy ≤ 2 weeks
  * TKI ≤ 2 weeks
  * Any experimental therapy ≤ 3 weeks or 5 half-lives, whichever is longer
  * Radiotherapy-wide therapy ≤ 3 weeks
  * Radiotherapy limited field (including stereotactic brain) ≤ 2 weeks
  * Antibody ≤ 3 weeks
* Any brain lesion requiring immediate local therapy
* Ongoing use of corticosteroids for central nervous system (CNS) symptoms at a dose of > 2 mg daily of dexamethasone (or equivalent)
* Leptomeningeal disease
* Uncontrolled seizures
* Participants for any chemotherapy cohort: ongoing Grade 2 or higher neuropathy of any cause
* Inability to swallow pills or any significant gastrointestinal disease that would preclude adequate oral absorption of medications.
* Ongoing adverse effects from prior treatment > CTCAE Grade 1 except for Grade 2 alopecia
* Corrected QT interval (QTc) of >470 milliseconds (ms) for females or >450 ms for males

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs; Phase 1a only) | 21 days
  DLTs will be used to support that the recommended doses for expansion are </= maximum tolerated dose (MTD)
Incidence of adverse events (AEs) | 24 months
  AEs will be used to support that the recommended doses for expansion are likely to be tolerable
Incidence of laboratory abnormalities | 24 months
  Clinically significant laboratory abnormalities will be used to support that the recommended doses for expansion are likely to be tolerable
Incidence of electrocardiogram abnormalities | 24 months
  Clinically significant electrocardiogram abnormalities will be used to support that the recommended doses for expansion are likely to be tolerable

SECONDARY OUTCOMES:
PK parameter of area under the curve of ELVN-002 (Phase 1a only) | 24 months
  The concentration of ELVN-002 measured in the blood over 24 hours at steady state
PK parameter of maximum concentration of ELVN-002 (Phase 1a only) | 24 months
  The maximum concentration of ELVN-002 measured in the blood at any time point at steady state
PK parameter of minimum concentration of ELVN-002 (Phase 1a only) | 24 months
  The minimum concentration of ELVN-002 measured in the blood at any time point at steady
PK parameter of terminal half life of ELVN-002 (Phase 1a only) | 24 months
  The half life of ELVN-002 calculated from the concentration of ELVN-002 measured in blood
Confirmed objective response rate (ORR) | 24 months
  For patients with measurable disease at baseline, confirmed response as assessed by investigator per RECIST v1.1
Duration of response (DOR; Phase 1b only) | 24 months
  The time from the first response to progression or death per RECIST v1.1
Brain metastases response (Phase 1b only) | 24 months
  For patients with measurable brain metastases at baseline, the percent of patients who have a confirmed response per RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (31):
- United States (3):
  - BRCR Medical Center Inc., Plantation, Florida
  - Washington University, St Louis, Missouri
  - NEXT Virginia, Fairfax, Virginia
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels
  - CHU de Liège, Liège
  - GZA Ziekenhuizen - Campus Sint-Augustinus, Wilrijk
- France (4):
  - Institut du Cancer de Montpellier - Val D'Aurelle, Montpellier
  - CHU de Poitiers, Poitiers
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Institut de Cancérologie Strasbourg Europe, Strasbourg
- Italy (6):
  - Azienda Ospedaliero-Universitaria Renato Dulbecco, Catanzaro
  - Istituto Europeo di Oncologia, Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda USL IRCCS di Reggio Emilia, Reggio Emilia
  - Fondazione Policlinico A. Gemelli IRCCS, Rome
- Radboud UMC, Nijmegen, Netherlands
- South Korea (5):
  - CHA Bundang Medical Center, Seongnam-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Soeul
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
- Spain (9):
  - NEXT Oncology-Hospital Quironsalud Barcelona, Barcelona
  - START Barcelona_HM Nou Delfos, Barcelona
  - Hospital Universitari Dexeus - Grupo Quironsalud, Barcelona
  - Instituto de Investigacion Oncologica Vall d'Hebron (VHIO) - EPON, Barcelona
  - Hospital Beata Maria Ana, Madrid
  - Clinica universitaria Navarra - Madrid, Madrid
  - START Madrid - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Clinica univeritaria Navarra - Pamplonas, Pamplona
  - Fundacion Instituto Valenciano de Oncologia, Valencia